CLINICAL TRIAL: NCT02783131
Title: Does Mednav, a Medical Navigation System, Aid Non-technical and Technical Skills in the Simulated Obstetric Emergency?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: C&W14/094
Record Dates: First submitted 2016-05-13; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Postpartum Hemorrhage,
Keywords: inventions; Simulation Training; Postpartum Haemorrhage; Non Technical Skills; teamwork; Crew Resource Management, Healthcare
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MedNav (Experimental): Team getting taught to use mednav, and using mednav in simulation managing Post partum Haemorrhage.
  Interventions: Device: MedNav
- non MedNav (No Intervention): Team undergoing routine simulation training in Post Partum Haemorrhage.

INTERVENTIONS:
Device: MedNav — MedNav is a tablet based platform device that acts to help teams manage emergencies. In the way that satellite navigation devices have replaced maps on journeys mednav has replaced paper based checklist and guidelines to give teams real-time guidance as the emergency happens. In supports teams by deligating, prompting and scribing as the emergency unfolds. The intervention arm will be taught how to use this device over 30 minutes and then use it in a simulated scenario managing a post partum haemorrhage.
  Other Names: A decision support tool
  Arms: MedNav

SUMMARY:
It is well known that medical errors account for a large amount of patient harm within the hospital setting. This is a significant problem within the emergency context. A system that acts as a prompt, guide and scribe for the obstetric emergency has been developed called 'Mednav'. Mednav is a navigation device for the management of medical emergencies; developed at Chelsea and Westminster Hospital since 2010. This is a device which acts similar to a satellite navigation devices in the automobile industry navigating you from A to B, MedNav navigates the clinician from the unwell patient to the well patient.

DETAILED DESCRIPTION:
Potential participants will be identified by those attending mandatory training/teaching. 2 weeks before their mandatory training they will be emailed with the study information leaflet and a link to a video which explains how to use Mednav. On the morning of the mandatory training/teaching they will be approached by the practice development midwife/Chief or Principle investigator who will give them a copy of the consent form and again the study information leaflet and show the Mednav video. Eligibility criteria will be checked and the study explained, before taking written informed consent.

Participants will personally sign and date the consent form, before any study specific procedures are performed.

Once the team is decided, the investigators will then randomise them to use of Mednav or no mednav, The participants will then undertake a simulated management of post partum haemorrhage which will be recorded for later review. Faculty will record the timing of completion of key technical skills.

A team of 8 assessors will review these simulated scenario recordings. Assessors will complete validated questionnaires to assess teamwork. Assessors will be asked to complete a technical skills list, showing timing and completion of various technical aspects of managing post partum Haemorrhage.

The end of the study will be when the required sample size has been recruited or significance found on interim data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Staff undertaking mandatory training at chelsea and westminster hospital

Exclusion Criteria:

* Non Consenting.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical Teamwork Scale | From date of randomisation to 72 weeks, each video will last 20 minutes. Assessors will review the videos at 12 weekly intervals at a sessions that last for up to 3 hours.
  A 15 point clinical teamwork scale that measures teamwork. This has separate points of: overall team work, communication, situation awareness, decision making, role responsibility, patient friendly. Scores for each section are between 0-10. 0 unacceptable, 1-3 Poor, 4-6 Average, 7-9 Good, 10 perfect. Validated for 3 assessors.
Global Assessment of Team Performance | From date of randomisation to 72 weeks, each video will last 20 minutes. Assessors will review the videos at 12 weekly intervals at a sessions that last for up to 3 hours.
  A 6 point scoring system with these subsections: Communication with patient and partner, Task management, Teamwork, Situational Awareness,Communication, Environment of Room. Each section is measured on a 5 point rating scale (1 poor performance, 5 excellent performance).
Technical Skill Achievement and timing | From date of randomisation to 72 weeks, each video will last 20 minutes. Assessors will review the videos at 12 weekly intervals at a sessions that last for up to 3 hours.
  A set of 11 key skills for managing a post partum haemorrhage. Massive obstetric haemorrhage call, Explore trauma, Palpate uterus, Examine placenta, IV Fluids started, Uterotonic started, Bloods taken and sent, Foley Cather inserted, Bimanual compression commenced, Blood transfusion commenced, Decision to move to theatre. Completion and time since emergency buzzer completion. This will be in the form of a table, which will include the skill and the time at which each skill is achieved. These timings will be recorded by the faculty of the simulation session.

SECONDARY OUTCOMES:
System Usability Score | From date of randomisation to 72 weeks, each simulation participant using mednav will answer the questionaire which will take 10 minutes.
  A validated usability score that gives results that can be interoperated into how 'usable' MedNav is.

CONTACTS AND LOCATIONS:
Overall Officials: shane p Duffy, MBCHB MRCOG, Study Director — Chelsea and Westminister NHS Foundation Trust